CLINICAL TRIAL: NCT00544219
Title: Prospective Evaluation of the Predictive Value of PET in Patients With Diffuse Large B-cell-lymphoma Under R-CHOP-14. A Multicenter Study
Brief Title: PET Scans in Patients With Diffuse Large B-Cell Lymphoma Receiving Rituximab, Cyclophosphamide, Doxorubicin, Vincristine, and Prednisone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 38/07; SWS-SAKK-38-07; EU-20763; EUDRACT-2007-001806-26; CDR0000569869
Record Dates: First submitted 2007-10-13; First posted 2007-10-16 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Lymphoma
Keywords: contiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; stage I adult diffuse large cell lymphoma; stage III adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; Cyclophosphamide; Doxorubicin; Prednisone; Vincristine; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- R-Chop 14 (Other): Standard treatment
  Interventions: Biological: rituximab; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: prednisone; Drug: vincristine sulfate; Procedure: positron emission tomography

INTERVENTIONS:
Biological: rituximab — 375 mg/m2 i.v. per cycle
  Other Names: Mabthera
Drug: cyclophosphamide — 750 mg/m2 i.v. per cycle
  Other Names: Endoxan
Drug: doxorubicin hydrochloride — 50 mg/m2 i.v. per cycle
  Other Names: Adriamycin, Adriblastin
Drug: prednisone — 100 mg/day p.o. per cycle
  Other Names: Deltasone, Orasone
Drug: vincristine sulfate — 1.4 mg/m2 (max. 2.0 mg) i.v. per cycle
  Other Names: Oncovin
Procedure: positron emission tomography — PET Scan during treatment

SUMMARY:
RATIONALE: Studying PET scans given to patients with cancer who are undergoing treatment may help doctors predict how patients will respond to treatment.

PURPOSE: This clinical trial is studying PET scans in patients with diffuse large B-cell lymphoma who are receiving rituximab together with cyclophosphamide, doxorubicin, vincristine, and prednisone.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate if an early positive positron emission tomography (PET) scan after 2 courses of rituximab with cyclophosphamide, doxorubicin hydrochloride, vincristine, and prednisone can be used to identify a group of patients having a poor prognosis.

Secondary

* To compare modified PET/CT scan response criteria with revised standard response criteria.
* To evaluate, in a prospective manner, whether a proliferation-inducing ligand (APRIL) expression is a prognostic factor in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive rituximab IV, cyclophosphamide IV, doxorubicin hydrochloride IV, and vincristine IV on day 1 and oral prednisone on days 1-5. Treatment repeats every 14 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Rituximab IV alone is continued for an additional 2 courses after completion of the initial 6 courses.

Patients undergo positron emission tomography (PET) scan prior to and after completion of study therapy. Patients also undergo PET scan after course 2, and those with a positive PET result undergo an additional PET scan after course 4.

Previously collected tumor samples are analyzed for a proliferation-inducing ligand (APRIL) expression.

After completion of study treatment, patients are followed periodically for up to 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion criteria:

* Histologically confirmed diagnosis of CD20+ diffuse large B-cell lymphoma (DLBCL)

  * Stage I-IV disease
  * All IPI risk groups
* Must be positron emission tomography (PET)-positive
* At least one measurable lesion ≥ 15 mm in its shortest axis (greatest transverse diameter) for jugulodigastric and infra-carinal lymph nodes with CT scan (MRI is allowed only if CT scan cannot be performed)

  * Otherwise the shortest axis (greatest transverse diameter) must be ≥ 10 mm
  * Lesions should be selected according to the following features:

    * Clearly measurable in two perpendicular dimensions
    * From as disparate regions of the body as possible
    * Include mediastinal and retroperitoneal areas of disease whenever these sites are involved

Exclusion criteria:

* Secondary DLBCL (in transformation)
* Evidence of symptomatic CNS disease

PATIENT CHARACTERISTICS:

Inclusion criteria:

* ECOG or WHO performance status 0-2
* Cardiac ejection fraction ≥ 50% as assessed by echocardiography
* Sufficient hematological values, hepatic and renal function
* Patient condition, compliance, and geographic proximity must allow proper staging and completion of treatment and follow-up
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 12 months after completion of study therapy

Exclusion criteria:

* Prior or concurrent hematological malignancies

  * Patients who have had prior solid organ tumors that required no treatment over the past 5 years and are currently disease-free are allowed
* Unstable cardiac disease within the past 6 months
* Any serious underlying medical condition (at the judgment of the investigator) that could impair the ability of the patient to participate in the study (e.g., active autoimmune disease, uncontrolled diabetes, HIV- and hepatitis-infection)
* Known hypersensitivity to any component of the study drugs

PRIOR CONCURRENT THERAPY:

Exclusion criteria:

* Prior chemotherapy, radiotherapy, or immunotherapy (e.g., rituximab) for lymphoma
* Prior anthracycline treatment
* Concurrent radiotherapy
* Concurrent regular corticosteroids in the past 4 weeks

  * Doses ≤ 20 mg/day of prednisone for indications other than lymphoma or lymphoma-related symptoms allowed
* Concurrent drugs contraindicated for use with the study drugs according to the Swissmedic-approved product information
* Other concurrent experimental drugs or other anticancer therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2007-09; Primary Completion 2012-09 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Event-free survival | at 2 years

SECONDARY OUTCOMES:
Event-free survival | at 5 years
Overall survival during follow-up | at 2 and 5 years
Objective response | at 2 years
Positron emission tomography (PET) results | at 2 years
Histological results of remaining PET-positive lesion(s) after treatment | at 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Mamot, MD, Study Chair — Kantonsspital Aarau; Mario Bargetzi, MD, Study Chair — Kantonsspital Aarau; Giovanni Martinelli, MD, Study Chair — European Institute of Oncology
Locations (19):
- European Institute of Oncology, Milan, Italy
- Switzerland (18):
  - Hirslanden Klinik Aarau, Aarau
  - Kantonspital Aarau, Aarau
  - Kantonsspital Baden, Baden
  - Praxis Dr. Streit, Baden
  - Saint Claraspital AG, Basel
  - Universitaetsspital-Basel, Basel
  - Oncology Institute of Southern Switzerland, Bellinzona
  - Inselspital Bern, Bern
  - Kantonsspital Bruderholz, Bruderholz
  - Kantonsspital Graubuenden, Chur
  - Hopital Cantonal Universitaire de Geneve, Geneva
  - Kantonsspital Liestal, Liestal
  - Kantonsspital Olten, Olten
  - Praxis Dr. Beretta, Rheinfelden
  - Kantonsspital - St. Gallen, Sankt Gallen
  - Regionalspital, Thun
  - Kantonsspital Winterthur, Winterthur
  - UniversitaetsSpital Zuerich, Zurich

REFERENCES:
- [Result] Juskevicius D, Jucker D, Klingbiel D, Mamot C, Dirnhofer S, Tzankov A. Mutations of CREBBP and SOCS1 are independent prognostic factors in diffuse large B cell lymphoma: mutational analysis of the SAKK 38/07 prospective clinical trial cohort. J Hematol Oncol. 2017 Mar 17;10(1):70. doi: 10.1186/s13045-017-0438-7. PMID 28302137
- [Result] Mamot C, Klingbiel D, Hitz F, Renner C, Pabst T, Driessen C, Mey U, Pless M, Bargetzi M, Krasniqi F, Gigli F, Hany T, Samarin A, Biaggi C, Rusterholz C, Dirnhofer S, Zucca E, Martinelli G. Final Results of a Prospective Evaluation of the Predictive Value of Interim Positron Emission Tomography in Patients With Diffuse Large B-Cell Lymphoma Treated With R-CHOP-14 (SAKK 38/07). J Clin Oncol. 2015 Aug 10;33(23):2523-9. doi: 10.1200/JCO.2014.58.9846. Epub 2015 Jul 6. PMID 26150440
- [Result] Tzankov A, Leu N, Muenst S, Juskevicius D, Klingbiel D, Mamot C, Dirnhofer S. Multiparameter analysis of homogeneously R-CHOP-treated diffuse large B cell lymphomas identifies CD5 and FOXP1 as relevant prognostic biomarkers: report of the prospective SAKK 38/07 study. J Hematol Oncol. 2015 Jun 14;8:70. doi: 10.1186/s13045-015-0168-7. PMID 26071053
- [Derived] Mendeville MS, Janssen J, Los-de Vries GT, van Dijk E, Richter J, Nijland M, Roemer MGM, Stathi P, Hijmering NJ, Bladergroen R, Pelaz DA, Diepstra A, Eertink CJ, Burggraaff CN, Kim Y, Lugtenburg PJ, van den Berg A, Tzankov A, Dirnhofer S, Duhrsen U, Huttmann A, Klapper W, Zijlstra JM, Ylstra B, de Jong D. Integrating genetic subtypes with PET scan monitoring to predict outcome in diffuse large B-cell lymphoma. Nat Commun. 2025 Jan 2;16(1):109. doi: 10.1038/s41467-024-55614-y. PMID 39747123
- [Derived] Ceriani L, Gritti G, Cascione L, Pirosa MC, Polino A, Ruberto T, Stathis A, Bruno A, Moccia AA, Giovanella L, Hayoz S, Schar S, Dirnhofer S, Rambaldi A, Martinelli G, Mamot C, Zucca E. SAKK38/07 study: integration of baseline metabolic heterogeneity and metabolic tumor volume in DLBCL prognostic model. Blood Adv. 2020 Mar 24;4(6):1082-1092. doi: 10.1182/bloodadvances.2019001201. PMID 32196557